CLINICAL TRIAL: NCT01126008
Title: A Phase II Trial of Concurrent Chemoradiotherapy With Weekly Docetaxel and Cisplatin for Locally Advanced Head and Neck Cancer
Brief Title: Concomitant Chemoradiotherapy (CCRT) With Weekly Docetaxel and Cisplatin for Locally Advanced Head and Neck Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Samsung Medical Center (Other)
Responsible Party: Principal Investigator, Keunchil Park, Principal investigator, Samsung Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2009-10-007
Record Dates: First submitted 2010-05-17; First posted 2010-05-19 (Estimated); Last update posted 2021-03-22 (Actual); Status verified 2021-03

CONDITIONS: Head and Neck Cancer
Keywords: locally advanced Squamous cell carcinoma
MeSH Terms: conditions — Head and Neck Neoplasms | interventions — Cisplatin

ARMS (1):
- weekly docetaxel and cisplatin (Experimental)
  Interventions: Drug: CCRT with weekly docetaxel & cisplatin

INTERVENTIONS:
Drug: CCRT with weekly docetaxel & cisplatin — radiotherapy: 70Gy/35 fraction for 7 weeks chemotherapy: docetaxel 20mg/m2 and cisplatin 20mg/m2 weekly for 6 weeks

SUMMARY:
This phase II trial is evaluating the efficacy of concurrent chemoradiation therapy with weekly docetaxel and cisplatin combination regimen.

DETAILED DESCRIPTION:
Many studies have shown the superiority of concurrent chemoradiotherapy over radiotherapy only in locally advanced head and neck cancer. Concurrent chemoradiotherapy with high dose cisplatin has been universally used regimen. In a large-scaled phase II trial, however, conducted by the European Organization for the Research and Treatment of Cancer (EORTC), docetaxel (100mg/m2) plus cisplatin (75mg/ m2) every three weeks regimen produced improved survival, nonetheless there was significant limitation to deliver full doses of treatment due to significant hematologic and non-hematologic toxicities. Previously, we showed the safety of the combination regimen of weekly docetaxel and cisplatin in concurrent chemoradiation treatment in a phase I study. We determined the MTD of docetaxel to be 20mg/m2 weekly when concurrently administered with conventional fractionation RT and weekly 20mg/m2 of cisplatin.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically confirmed squamous cell carcinoma of the head and neck (SCCHN) of one of following sites : oral cavity, oropharynx, larynx, or hypopharynx
2. Unresectable Stage III - ⅣB disease
3. previously untreated for head & Neck cancer with chemotherapy or radiotherapy
4. 18 and over
5. Performance status ECOG 0-1
6. Absolute neutrophil count ≥ 1,500/mm3
7. Platelet count ≥ 75,000/mm3
8. Hemoglobin > 9.0 g/dL
9. Bilirubin ≤ 1.5 times upper limit of normal (ULN)
10. AST or ALT, and alkaline phosphatase meeting 1 of the following parameters:Alkaline phosphatase ≤ 1.5 times ULN AND AST or ALT ≤ 5 times ULN Alkaline phosphatase ≤ 2.5 times ULN AND AST or ALT ≤ 1.5 times ULN Alkaline phosphatase ≤ 5 times ULN AND AST or ALT ≤ ULN
11. serum creatinine ≤ 1.5 mg/dl or creatinine clearance ≥ 60 ml/min

Exclusion Criteria:

1. Distant metastatic disease (M1)
2. Prior chemotherapy or RT for Head and neck cancer
3. Synchronous or concurrent head and neck primary tumors
4. Lip, nasopharynx, nasal cavity, salivary gland, or sinuses
5. No other invasive malignancy within the past 3 years except nonmelanoma skin cancer or papillary thyroid cancer
6. Other concurrent illness that would preclude study participation
7. Other concurrent physical condition (e.g., infectious disease) that would preclude study participation
8. pregnant or nursing
9. Fertile patients must use effective contraception during and for 3 months after study participation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2009-11-16 (Actual); Primary Completion 2016-04-15 (Actual); Study Completion 2016-04-15 (Actual)

PRIMARY OUTCOMES:
Complete response rate | 3-4 weeks after completion of CCRT

SECONDARY OUTCOMES:
quality of life | Pretreatment & 3-4 weeks after completion of treatment
overall survival rate | 2 year
disease free survival rate | 2 year

CONTACTS AND LOCATIONS:
Locations (1):
- Samsung Medical Center, Seoul, South Korea